CLINICAL TRIAL: NCT07237607
Title: Developing an Artificial Intelligence (AI)-Powered Exposure Therapy Chatbot for Adolescents and Young Adults With Eating Disorders
Brief Title: Developing an Artificial Intelligence (AI) Chatbot for Adolescents and Young Adults With Eating Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Jamal Essayli, Assistant Professor, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26987
Record Dates: First submitted 2025-11-14; First posted 2025-11-20 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- "Exp-ED" Digital Exposure-Therapy Chatbot app (Experimental): Exp-ED will target anxiety about weight gain through an exposure based treatment.
  Interventions: Device: "Exp-ED" Digital Exposure-Therapy Chatbot app

INTERVENTIONS:
Device: "Exp-ED" Digital Exposure-Therapy Chatbot app — Exp-ED is a text-based digital health application designed for smartphones and personal computers. It provides exposure-based content to adolescents and young adults with eating disorders. The chatbot guides users through exposure exercises (structured steps to reduce anxiety over time), records subjective distress ratings (self-reported anxiety scores), and offers evidence-based coping prompts. These sessions are intended to supplement clinical care during a six-week partial hospitalization program.

SUMMARY:
The goal of this study is to develop and refine an artificial intelligence (AI)-powered Exposure Therapy for Eating Disorders chatbot web-app that effectively engages adolescents and young adults and decreases anxiety about weight gain. Participants will use the web-app as a supplemental therapeutic tool during their first six weeks of treatment in a Partial Hospitalization Program. Participants will complete assessments every two weeks, including: (1) semi-structured interviews about their experience with the chatbot web-app; (2) implementation outcome measures (e.g., feasibility, usability, acceptability); and (3) anxiety about weight gain.

DETAILED DESCRIPTION:
The overarching goal of this study is to develop and refine an AI-powered Exposure Therapy for Eating Disorders (Exp-ED) chatbot app that effectively engages adolescents and young adults (AYAs) with eating disorders (EDs) and decreases anxiety about weight gain. The investigators will enroll 20 AYAs (ages 12-26 years) entering the Partial Hospitalization Program (PHP) for EDs at the Penn State Milton S. Hershey Medical Center. The initial version of the Exp-ED chatbot app will be developed by an interdisciplinary team with expertise in exposure therapy for EDs (Dr. Essayli), AI (Dr. Nawab), and implementation science (Dr. Lenker). Participants will use the Exp-ED chatbot app as a supplemental therapeutic tool during their first six weeks of PHP treatment. Participants will complete assessments every two weeks, including: (1) semi-structured interviews about their experience with the Exp-ED chatbot app, including design issues and engagement barriers; (2) implementation outcome measures (e.g., feasibility, usability, acceptability); and (3) anxiety about weight gain. Success will be evaluated using pre-determined benchmarks derived from previous mental health chatbot research. This project has two aims:

Aim 1: Iteratively adapt an exposure therapy chatbot app for AYAs with EDs. The investigators will conduct monthly reviews of mixed-methods data and use the Framework for Reporting Adaptations and Modifications-Enhanced (FRAME) to systematically document and evaluate modifications to the chatbot app. Each revised version will be tested with new participants, creating an iterative development process that continues throughout the project period. All adaptation decisions and their empirical foundations will be documented to create a comprehensive record of the app's development via implementation science frameworks.

Aim 2. Evaluate the feasibility, usability, acceptability, and preliminary efficacy of the Exp-ED chatbot app. H2.1: The investigators will recruit ≥50% of eligible AYAs with EDs. H2.2: Over the six-week project period, participants will use the app ≥18 times. H2.3: Participants will engage with the chatbot for ≥100 minutes total. H2.4: Participants will rate the Exp-ED chatbot app as acceptable (score ≥68 on the System Usability Scale). H2.5: Participants will report a ≥50% reduction in anxiety about weight gain.

ELIGIBILITY:
Inclusion Criteria:

* Age is between or equal to 12-26 years
* Admitted to the Penn State Health Eating Disorder Partial Hospital Program (PHP) or Intensive Outpatient Program (IOP)
* Have a personal smartphone
* Have a diagnosis of anorexia nervosa (AN), bulimia nervosa (BN), binge-eating disorder (BED), or other specified feeding or eating disorder (OSFED)
* Be English speaking

Exclusion Criteria:

* Diagnosis of avoidant/restrictive food intake disorder (ARFID)
* Have acute suicidality
* Diagnosis of an intellectual disability

Ages: 12 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of times participants use web-app. | End of Week 2, End of Week 4, End-of-Treatment (Week 6)
  The investigators will measure the number of times participants use the web-app
Number of minutes participants engage with the web-app. | End of Week 2, End of Week 4, End-of-Treatment (Week 6)
  The investigators will measure the number of minutes participants engage with the web-app
Percent of eligible Adolescents and Young Adults Consented | Through study completion, an average of 1 year
  The investigators will measure the percent of eligible adolescents and young adults who consent to the study.
System Usability Scale Survey (SUS) | End of Week 2, End of Week 4, End-of-Treatment (Week 6)
  The System Usability Scale Survey (SUS) is a 10-item self-report questionnaire that examines the participant's attitude towards the web-app. Scores range from 10-50, with higher scores indicating a better overall experience with the app.
Weight Gain Anxiety Questionnaire | Baseline, End of Week 2, End of Week 4, End-of-Treatment (Week 6)
  The Weight Gain Anxiety Questionnaire is a 12-item self-report questionnaire that targets anxiety about weight gain. The scores are measured on a 0-100 scale, with the higher the score indicating more distress about weight gain, with the exception for question 12 which is reverse scored.

SECONDARY OUTCOMES:
Clinical Impairment Assessment (CIA) | Baseline, End-of-Treatment (Week 6)
  The Clinical Impairment Assessment Questionnaire (CIA) is a 16-item self-report measure of the severity of psychosocial impairment due to eating disorder features and focuses on the past 28 days. The 16 items cover impairment in domains of life that are typically affected by eating disorder psychopathology: mood and self-perception, cognitive functioning, interpersonal functioning, and work performance. The responses are scored 0,1,2 and 3, with a higher rating indicating a higher level of impairment. The total range is between 0 and 48.
Eating Disorder Examination - Self-Report Questionnaire (EDE-Q) | Baseline, End-of-Treatment (Week 6)
  The Eating Disorder Examination Questionnaire (EDE-Q) is a 28-item self-report questionnaire. It was designed to assess the range, frequency, and severity of behaviors associated with a diagnosis of an eating disorder. A global score is obtained by summing the four subscales scores (ranging from 0-6) and dividing the total by the number of subscales (4). The score of items are calculated and range from 0 to 6. The higher score indicate greater ED symptoms.
Eating Disorder Fear Questionnaire (EDFQ) | Baseline, End-of-Treatment (Week 6)
  The Eating Disorder Fear Questionnaire (EDFQ) is a 20-item self-report questionnaire. It examines the participant's severity of behaviors associated with a diagnosis of an eating disorder. The response range between 1 to 7 with a total range of 20 to 140. The higher rating indicates a higher severe impairment.
Fear of Food Measure (FOFM) | Baseline, End-of-Treatment (Week 6)
  The Fear of Food Measure (FORM) is a 23-item self-report questionnaire. It examines the participant's severity of behaviors associated with a diagnosis of an eating disorder. Each item is scored on a 1-7 scale. The questionnaire range from 23 to 161 meaning 23: no fear of food and 161 meaning severe fear of food.
Generalized Anxiety Disorder-7 (GAD-7) | Baseline, End-of-Treatment (Week 6)
  The Generalized Anxiety Disorder-7 is a 7-item self-report questionnaire that targets anxiety symptoms. The scores range from 0 to 21, with higher scores indicating higher levels of anxiety.
Patient Health Questionnaire-9 (PHQ-9) | Baseline, End-of-Treatment (Week 6)
  The Patient Health Questionnaire-9 is a 9-item self-report questionnaire that targets depressive symptoms. The scores range from 0-27, with higher scores indicating a higher level of depression.
Eating Anxiety Questionnaire | Baseline, End of Week 2, End of Week 4, End-of-Treatment (Week 6)
  The Eating Gain Anxiety Questionnaire is a 14-item self-report questionnaire that targets anxiety about eating fear foods. The scores are measured on a 0-100 scale, with the higher the score indicating more distress about eating fear foods, with the exception for question 12 which is reverse scored.

OTHER OUTCOMES:
Columbia Suicide Severity Rating Scale (CSSRS) | Baseline
  Evidence-based metric evaluating for presence of suicidal ideation and severity. Scores range from 1 (low risk) to 3 (high risk).